CLINICAL TRIAL: NCT01540552
Title: Evolution of Undetermined Ld-CT Detected Lung Nodules Among a Randomized Phase II Trial With Inhaled Budesonide
Brief Title: Natural History of Lung Nodules Seen on CT Scans From Participants at High-Risk of Developing Lung Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA11-1128; MDA-MDA05-5-03; CDR0000726610 (Other: NCI Clinical Trials)
Record Dates: First submitted 2012-02-22; First posted 2012-02-29 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer; Precancerous Condition
Keywords: lung cancer; precancerous condition; lung nodules; CT Scan
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions | interventions — Diagnosis, Computer-Assisted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Budesonide Arm: Retrospective Medical Chart Review of low dose CT scans for participants who received Budesonide.
  Interventions: Other: medical chart review; Procedure: computed tomography; Procedure: computer-aided detection/diagnosis
- Placebo Arm: Retrospective Medical Chart Review of low dose CT scans for participants who received Placebo.
  Interventions: Other: medical chart review; Procedure: computed tomography; Procedure: computer-aided detection/diagnosis

INTERVENTIONS:
Other: medical chart review
Procedure: computed tomography
Procedure: computer-aided detection/diagnosis

SUMMARY:
RATIONALE: Comparing lung CT scans from participants with lung nodules at high-risk for lung cancer may help doctors learn more about the disease and find better methods of treatment.

PURPOSE: This trial studies the natural history of lung nodules using CT scans from participants at high-risk for lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluation of lung nodules (target and non-target lesions) detected during annual low-dose (ld) computed tomography (CT) scans and measured for three years after study completion in subjects enrolled in a randomized, phase IIb, placebo-controlled trial with inhaled budesonide (both person-specific and lesion-specific analyses will be performed).

Secondary

* Lung cancer detection rate in the two arms.
* Appearance of new nodules in the two arms.

OUTLINE: Low-dose CT scans are analyzed retrospectively for the natural progression of undetermined lung nodules. Nodule dimension will be evaluated according to maximum diameter and volume, when feasible. Volume measurements are performed using an automatic and semi-automatic computer-aided diagnosis (CAD) system. Lesion-specific and person-specific analysis are performed by measure of average change in size of the target lesions or number of lesions.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Annual Computed Tomography (CT) scans obtained from participants with undetermined lung nodules detected by low-dose CT enrolled in both of the following trials:

  * A large-scale COSMOS screening trial

    * Three annual CT scans obtained as part of the COSMOS trial after budesonide study treatment completion
  * The MDA05-5-01, a subset of COSMOS trial participants, a randomized phase II trial of inhaled budesonide twice daily versus placebo

    * Two CT scans performed as part of the budesonide protocol (MDA05-5-01)
* Only CT scans from participants enrolled in both trials will be used

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants previously enrolled in two trials: (1) a large scale COSMOS trial and (2) a subset of the COSMOS trial (MDA05-5-01 Budesonide study and treated for one year). Only participants enrolled in both trials will be included.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Natural evolution of lung nodules | 5 year review period

SECONDARY OUTCOMES:
Lung cancer detection rate | 5 year review period
Appearance of new nodules | 5 year review period

CONTACTS AND LOCATIONS:
Overall Officials: Powel H. Brown, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Veronesi G, Lazzeroni M, Szabo E, Brown PH, DeCensi A, Guerrieri-Gonzaga A, Bellomi M, Radice D, Grimaldi MC, Spaggiari L, Bonanni B. Long-term effects of inhaled budesonide on screening-detected lung nodules. Ann Oncol. 2015 May;26(5):1025-1030. doi: 10.1093/annonc/mdv064. Epub 2015 Feb 11. PMID 25672894
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org